CLINICAL TRIAL: NCT07206355
Title: In-Depth Characterisation of Biliary Strictures and Hepato-Pancreato-Biliary Focal Lesions for Development of New Technologies to Tackle Hepato-Pancreato-Biliary Cancers
Acronym: Map HPB
Status: Not yet recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 25014
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-07

CONDITIONS: Biliary Tract Cancer (BTC); Biliary Tract Cancer (CCA); Cholangiocarcinoma; Cholangiocarcinoma Cancer; Cholangio Carcinoma; Pancreatic Cancer; Pancreatic Cyst
Keywords: biliary tract cancer; Pancreatic Cancer; Pancreatic Cyst; Pancreatic lesions; Biliary Tract Cancer (BTC); Cholangiocarcinoma
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma; Pancreatic Neoplasms; Pancreatic Cyst

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Biospecimen including tissue, body fluids (bile, pancreatic cyst fluid, blood) will be collected either through the standard care pathway or during regular clinical appointments. Blood samples from the patients will be collected at the time of enrolment to the study and at follow up visits. We will try to collect samples (extra 3 vials up to 20 ml) when blood samples are collected for clinical tests.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients undergoing investigations for the diagnosis and treatment of a HPB focal lesions: (a) (up to 140 cases) Patients undergoing investigations for the diagnosis and treatment of a HPB focal lesions (in the liver, gall bladder, bile duct, biliary tract or pancreas), including stricture and pancreatic cysts. Investigations will be determined and performed as a part of the standard of care. (The type of investigations varies and is decided by the clinician in charge or multidisciplinary team meeting decision.) These will be performed using either endoscopic or radiologic approaches including:
  * Endoscopic Ultrasound (EUS) with endoscopic fine needle acquisition of tissue (FNA/FNB/cyst wall biopsy) for pancreatic cysts or any pancreatic lesion, Endoscopic retrograde cholangio-pancreatography (ERCP) and/or cholangioscopy (SpyGlass™ device) for liver or biliary strictures.
  * Percutaneous sampling of liver or biliary strictures using ultrasound or percutaneous transhepatic cholangiography (PTC) and/or SpyGlass Discover™ cholangioscopy.
- b. Patients undergoing surgical resection: (up to 20 cases) Patients undergoing surgical resection (of liver, pancreas, gallbladder or bile duct) as standard of care for any underlying condition.

SUMMARY:
Hepato-Pancreato-Biliary (HPB) cancers originating in the liver, bile ducts, pancreas, and gall bladder represent a rising global health challenge, with incidence doubling in the UK over the past decade. Cholangiocarcinoma (CCA) and pancreatic cancer are particularly aggressive, often detected late due to non-specific symptoms and difficulties in sampling or imaging. In the UK, CCA affects around 3,000 people annually, with only 13% surviving 3 years, while pancreatic cancer has a 5-year survival of 8.3%. Diagnosis is complicated by the anatomical narrowness of the bile duct and the similarity between malignant and benign strictures. Standard imaging often cannot distinguish between inflammation and cancer, while tissue sampling is challenging, paucicellular, and limited in sensitivity, necessitating repeated biopsies. Yet, accurate characterisation is critical as NICE now recommends targeted therapies (FGFR2, NTRK, MSI-H/dMMR, IDH1 mutations) that require molecular profiling.

Both CCA and PDAC display high heterogeneity, further complicating treatment. Emerging approaches such as Raman spectroscopy can map malignant tissues by detecting vibrational energy shifts, but require further validation due to weak signals. For focal or cystic HPB lesions not well visualised by conventional imaging, novel modalities like ultra-thin endoscopes with scattering/absorption imaging are being developed for improved early diagnosis.

Management of biliary obstruction frequently involves stenting to restore bile flow, essential for palliation and pre-treatment optimization. However, stent failure from tumour ingrowth, displacement, or erosion remains common, and evidence for best stent use is limited. Novel approaches, including drug-eluting coatings and nanoparticle-mediated wireless treatment delivery, are being investigated.

To overcome diagnostic and therapeutic barriers, flexible snake-like robotic systems with navigation, sampling, spectroscopy, and treatment capabilities are being developed. These devices, alongside ultra-thin endoscopes and integrated Raman spectroscopy, aim to characterise strictures, generate 3D imaging in ex-vivo HPB tissue, and permit targeted ablation. Parallel work will explore molecular and fluid-based biomarkers (blood, bile, cyst fluid) to support minimally invasive diagnosis and monitoring.

Through integration of engineering, molecular diagnostics, and device innovation, this transdisciplinary research programme (UKRI and MRC funded) seeks to transform early detection, accurate diagnosis, and novel treatment of HPB cancers, thereby improving outcomes in CCA, pancreatic malignancy, and other clinically similar biliary disorders.

Aim:

To provide a detailed understanding of the characteristics (including clinical and molecular) of liver and pancreatic biliary focal lesions (inflammatory and cancerous) and create a bioresource of liver, pancreas, gallbladder and biliary tract associated tissue and fluids (biopsies, brushings, resected tissues, bile and cyst fluid and blood samples) in order to develop innovative tools for accurate diagnosis and treatment.

Study Configuration: Prospective Longitudinal Cohort study Setting: Secondary care centre, Nottingham University Hospitals NHS Trust. (NUH).

Co-ordinated by the NIHR Nottingham Biomedical Research Centre Description of interventions: This is an observational study involving collecting tissue or body fluids (such as bile or pancreatic cyst fluid) during clinical care in addition to collection of blood samples (for DNA, serum and plasma) and data collection.

Surplus tissue residual to the requirements for standard care will be stored and used. Additional tissue samples and body fluid samples collected for research at time of clinical investigations will not be increasing the risk of the clinical procedure.

Blood samples will be collected from patients at the time of enrolment in the study. These may be collected before and/ or after diagnosis is secured.

Duration of study: Overall duration: 60 months Outcome measures: - To report the proportion of patients where adequate tissue could be retrieved from HPB biopsy to come to definitive diagnosis using standard of care.

* To report the proportion of patients where adequate tissue could be retrieved from biopsy to perform molecular characterisation of HPB samples, beyond standard cyto/histology, using advanced optical-spatial technologies currently under development.
* To report the proportion of patients where definitive diagnosis of mucinous cystic neoplasm could be made in patients with pancreatic cyst using standard care
* To report the proportion of patients where molecular characterisation beyond standard cyto/histology could be made in patients with pancreatic cyst using exploratory new technologies under development through ex-vivo experiments
* To report the correlation between Raman Spectroscopy and standard cyto/histology for identification of cancer in HPB samples

ELIGIBILITY:
Inclusion Criteria:

* Aged 16 years and over
* Ability to provide informed consent to participate in the study
* Patients attending Nottingham University Hospitals NHS Trust (NUH) as part of standard clinical care for either:

  * the diagnosis and treatment of suspected biliary stricture or any focal lesion in the Hepato-Pancreato-Biliary (HPB) tract (clinically / radiologically) including liver or pancreatic lesion or pancreatic cyst
  * surgical resection treatment of liver, pancreas, or gall bladder including Whipple Procedure (pancreaticoduodenectomy surgery), gall bladder resection (cholecystectomy), hepatic resection

Exclusion Criteria: No exclusion criteria

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing investigations for the diagnosis and treatment of a HPB focal lesions Patients undergoing surgical resection (of liver, pancreas, gallbladder or bile duct)
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
To characterise biliary strictures and hepato-pancreato-biliary (HPB) focal lesions | 3 years
  To characterise biliary strictures and hepato-pancreato-biliary (HPB) focal lesions to diagnose cancers including cholangiocarcinoma (CCA) in a prospective patient cohort, establishing clinical features (manifestations, pathology, cytology, treatment responses and outcomes) and molecular, cellular, structural and physical properties.

SECONDARY OUTCOMES:
To create a database and associated bioresource of HPB tissues | 3 years
  To create a database and associated bioresource of HPB tissues (, including the liver, bile duct, gallbladder and pancreas), with or without any focal lesion, for analysis of diagnostic and treatment technologies under development in the laboratory (super-slender robot, ultra-thin scattering absorption and shape endoscope, and electrical actuation technology).
To develop a library of images | 3 years
  To develop a library of images (Endoscopic, Radiology, Raman Spectroscopy) of biliary strictures and HPB lesions or HPB resected tissue linked to specific cyto/ histology and molecular information.
To correlate Raman Spectroscopic images | 3 years
  To correlate Raman Spectroscopic images with molecular characteristics of the HPB samples.
To identify genetic markers and biomarkers for early diagnosis | 3 years
  To identify genetic markers and biomarkers for early diagnosis and monitoring of HPB lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Guruprasad P Aithal, MBBS, MD, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No